CLINICAL TRIAL: NCT04962074
Title: Sperm Selection and Embryo Development: Comparison of the Density Gradient Centrifugation and Microfluidic Chip Sperm Preparation Methods
Brief Title: Sperm Selection and Embryo Development: Comparison of the Density Gradient Centrifugation and Microfluidic Chip Sperm Preparation Methods Sperm Selection and Embryo Development: Comparison of the Density Gradient Centrifugation and Microfluidic Chip Sperm Preparation Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019
Record Dates: First submitted 2021-06-25; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Reduced Sperm Motility; IVF; ICSI; Astheno Teratozoospermia
Keywords: Sperm; IVF; ICSI; Abnormal morphology of sperm; Astheno Teratozoospermia; Microfluidic chip
MeSH Terms: conditions — Asthenozoospermia | interventions — Centrifugation, Density Gradient

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Density gradient method (Experimental): Sperm prepared by density gradient method
  Interventions: Device: Density gradient
- Microfluidic chip (Experimental): Sperm prepared by microfluidic chip method
  Interventions: Device: Microfluidic sperm sorting chip

INTERVENTIONS:
Device: Microfluidic sperm sorting chip — Fertile Ultimate® (Koek Biotechnology, Turkey) microfluidic sperm sorting chips
  Arms: Microfluidic chip
Device: Density gradient — Density gradient centrifugation
  Arms: Density gradient method

SUMMARY:
Purpose: To compare the effects of the density gradient centrifugation and microfluidic chip sperm preparation methods on embryo development in a study population with astheno-teratozoospermia.

Materials and Methods: In this prospective study, the semen samples of the patients with astheno-teratozoospermia were divided into two groups for preparation with either the microfluidic or density gradient methods. Selected spermatozoa were used to fertilize the mature sibling oocytes. Semen parameters and embryo development on days 3 and 5 were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Infertile men with astheno-teratozoospermia
* Women were aged from 18 to 39
* Women had at least two mature oocytes.

Exclusion Criteria:

* MI oocytes

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Split semen samples from the same population of infertile men with astheno-teratozoospermia were used to fertilize the mature sibling oocytes.
Enrollment: 22 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Semen parameters after sperm preparation with either method: semen volume | up to 7 months
  semen volume (ml)
Semen parameters after sperm preparation with either method: sperm concentration | up to 7 months
  sperm concentration (106/ml)
Semen parameters after sperm preparation with either method: total motility | up to 7 months
  total motility (%)
Semen parameters after sperm preparation with either method: progressive motility | up to 7 months
  progressive motility (%)
Embryo development after sperm preparation with either method | up to 7 months
  Embryo development and blastocyst formation were evaluated on days 1, 3 and 5 based on the criteria reported by Veeck and Zaninovic, 2003

CONTACTS AND LOCATIONS:
Locations (1):
- MaltepeU, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No